CLINICAL TRIAL: NCT07129057
Title: Effect of Mindfulness-Based Protocols on Psychological Parameters and Biological Markers in Populations Exposed to Conditions of Persistent Distress: a Randomized Controlled Trial in Healthcare Workers
Brief Title: Effect of Mindfulness-Based Protocols on Psychological Parameters and Biological Markers in Populations Exposed to Conditions of Persistent Distress
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda Unita Sanitaria Locale di Piacenza (Other)
Collaborators: University of Siena, Italy (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MINDFULNESS-BASED
Record Dates: First submitted 2025-07-25; First posted 2025-08-19 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Distress, Psychological
Keywords: Attention and awareness; Clinical psychology; Mindfulness; Randomized Controlled Trial; Stress biomarkers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MBSR program (Experimental): The MBSR program is an introductory course to mindfulness practices that operate through the systematic and continuous cultivation of specific mental states that promote a different relationship with stress and discomfort.
  Interventions: Other: MBSR program
- Control (No Intervention): No attending to the MBSR program

INTERVENTIONS:
Other: MBSR program — The MBSR program lasts eight consecutive weeks (two months), with group sessions lasting two and a half hours each and an intensive 8-hour full-day practice session. At each session, the participants receive audio tracks for daily home practice.
  Arms: MBSR program

SUMMARY:
The goal of this clinical trial is to learn if a Mindfulness-Based Stress Reduction (MBSR) training can improve the mental health and well-being of healthcare professionals (HCPs) exposed to prolonged severe stress conditions.

The main questions it aims to answer are:

* Does an 8-week MBSR training lower the cortisol levels of HCPs exposed to prolonged severe stress conditions?
* Does an 8-week MBSR training modify the psychological condition of HCPs exposed to prolonged severe stress conditions? Researchers will compare an 8-week MBSR training to no-training to see if MBSR training works to improve the mental health and well-being of HCPs.

Participants will:

* Partecipate or not partecipate to the MBSR training for 8 weeks
* Visit the clinic at baseline, after the 8-week intervention (T1), and at follow-up after 6 months for checkups and tests

ELIGIBILITY:
Inclusion Criteria:

* Healthcare workers belonging to the Dept. of Mental Health, Onco-hematology, Medicine, and Intensive Care, who are frequently exposed to situations of severe and prolonged stress
* age between 18 and 65 years
* informed consent

Exclusion Criteria:

* Use of psychotropic drugs in the previous 2 months
* Previous mindfulness training
* Medical conditions preventing participation in group sessions
* Current pregnancy.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2020-10-10 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
Cortisol level | At baseline before the intervention (T0), after the 8-week intervention (T1), and at follow-up after 6 months (T2)
  To assess cortisol levels, at baseline (T0), T1, and T2, saliva samples will be collected using Salivettes (Sarstedt) 30 minutes after waking up. Participants will be instructed not to drink, eat, chew gum, or brush their teeth in the 30 minutes preceding the sample collection. To collect the saliva, participants will be advised to rinse their mouth with water for 30 seconds, wait 10 minutes, and then remove the swab from the Salivette and chew it for about 2 minutes to stimulate salivation. The swab will be reinserted into the Salivette, frozen at -20°C and stored at the Laboratory of the AUSL Piacenza Centre. Then, sample will be shipped to the University of Siena for further analysis. Upon arrival at the laboratory, the samples will be thawed and centrifuged at 2000 × g for 5 minutes at 4°C. Salivary cortisol levels will be assayed by an Enzyme Immunoassay kit (Arbor Assays Inc., Ann Arbor, Michigan, USA).

SECONDARY OUTCOMES:
Psychometric evaluation of stress and burnout by Job Strain subscale of the Italian Cardiologists' Undetected Distress Study (IANUS) | At baseline before the intervention (T0), after the 8-week intervention (T1), and at follow-up after 6 months (T2)
  The IANUS consists of 15 items for measuring 4 main factors. Items are scored on a Likert-type response scale (never=1; sometimes=2; often=3; almost always=4). The score of the Job Strain 5-item subscale ranges from 0 to 100 [sum of item scores *100/(4*5)], with higher values corresponding to greater job strain.
Psychometric evaluation of stress and burnout by Positive Meaning subscale of the Italian Cardiologists' Undetected Distress Study (IANUS) | At baseline before the intervention (T0), after the 8-week intervention (T1), and at follow-up after 6 months (T2)
  The IANUS consists of 15 items for measuring 4 main factors. Items are scored on a Likert-type response scale (never=1; sometimes=2; often=3; almost always=4). The score of the Positive Meaning 4-item subscale ranges from 0 to 100 [sum of item scores *100/(4*4)], with higher values corresponding to greater positive meaning of work by the partecipant.
Psychometric evaluation of stress and burnout by Emotional Fatigue subscale ofthe Italian Cardiologists' Undetected Distress Study (IANUS) | At baseline before the intervention (T0), after the 8-week intervention (T1), and at follow-up after 6 months (T2)
  The IANUS consists of 15 items for measuring 4 main factors. Items are scored on a Likert-type response scale (never=1; sometimes=2; often=3; almost always=4). The score of the Emotional Fatigue 3-item subscale ranges from 0 to 100 [sum of item scores *100/(4*3)], with higher values corresponding to greater emotional fatigue of the partecipant.
Psychometric evaluation of stress and burnout by Relational Difficulty subscale of the Italian Cardiologists' Undetected Distress Study (IANUS) | At baseline before the intervention (T0), after the 8-week intervention (T1), and at follow-up after 6 months (T2)
  The IANUS consists of 15 items for measuring 4 main factors. Items are scored on a Likert-type response scale (never=1; sometimes=2; often=3; almost always=4). The score of the Relational Difficulty 3-item subscale ranges from 0 to 100 [sum of item scores *100/(4*3)], with higher values corresponding to greater relational difficulties by the partecipant.
Psychometric evaluation of stress and burnout by the Perceived Stress Scale (PSS) | At baseline before the intervention (T0), after the 8-week intervention (T1), and at follow-up after 6 months (T2)
  The PSS measures the degree to which situations in a person's life are appraised as stressful. Each item was rated by the subject on a scale ranging from 0 (never) to 4 (very often). The scale values range from 0 to 40, with a higher score indicating a higher degree of subjective stress. Total scores 0-13 are considered low perceived stress, 14-26 as moderate perceived stress, and 27-40 as high perceived stress.
Psychometric evaluation of awareness and mindfulness skills by the Mindfulness Awareness Attention Scale (MAAS) | At baseline before the intervention (T0), after the 8-week intervention (T1), and at follow-up after 6 months (T2)
  The MAAS is a 15-item scale investigating awareness and attention to what is happening in the present. The MAAS is a 15-item self-report instrument designed to measure dispositional mindfulness, specifically the frequency of open or receptive attention to and awareness of present-moment experiences. Participants rate each item (e.g., "I find it difficult to stay focused on what's happening in the present") on a 6-point Likert scale ranging from 1 (almost always) to 6 (almost never), with higher scores indicating greater mindfulness. The MAAS has demonstrated high internal consistency and good psychometric properties in both clinical and non-clinical populations.
Psychometric evaluation of psychophysiological distress and quality of life by the Psychological General Well-Being Short (PGWB-S) | At baseline before the intervention (T0), after the 8-week intervention (T1), and at follow-up after 6 months (T2)
  PGWB-S is a 6-item, rated on a 6-point scale, health-related Quality of Life questionnaire derived from the 22-item Psychological General Well-Being Index, developed in the United States. It produces a self-perceived evaluation of psychological well-being expressed by a summary score, which reaches a maximum of 30 points, representing the best achievable "well being".
  The PGWB-S showed good acceptability and validity for use in various settings in Italy.

CONTACTS AND LOCATIONS:
Locations (1):
- Liaison Psychiatry and Social Inclusion Unit of the Local Health Unit ("Azienda Unità Sanitaria Locale", AUSL) of Piacenza, Piacenza, Italy

IPD SHARING:
Plan to Share IPD: No